CLINICAL TRIAL: NCT02628808
Title: Search of Susceptibility Genes in Autism Spectrum Disorders
Brief Title: Susceptibility Genes in Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C07-33; 2008-A00019-46 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-09-26; First posted 2015-12-11 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorders
Keywords: autism; asperger; Pervasive Developmental Disorder No Otherwise Specify; gene; polymorphism; mutation
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from subjects will be stored in the biobank of our study. From some patients with deleterious mutations in synaptic genes, cells (PBMC, Keratinocytes ou Fibroblasts) will be sampled from derivation in Induced Pluripotent Stem Cells.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Autism Spectrum Disorder: For all patients included in the study, core assessment carried out by either collaborating partners consists of diagnosis using the Autism Diagnostic Interview-Revised (ADI-R) criteria for autism and Autism Diagnostic Observation Schedule (ADOS-G) criteria for autism or Autism Spectrum Disorders. Patients with profound intellectual disability or with a known medical cause of autism, such as neurocutaneous syndromes, Fragile X, metabolic disorders, extreme prematurity, congenital rubella and other prenatal or postnatal neurological infections or gross dysmorphology, will be excluded.
- controls: Age 2 to 65 Healthy individuals with or without idiopathic surgical or urological conditions (e.g. orthopaedic conditions, hernia repairs, renal malformations, pre- or post-circumcision, phimosis, balanitis, scoliosis, congenital hip dislocation, adenoid or tonsil removal, dental procedures such as wisdom tooth extraction, cosmetic procedures such as removal of skin tags or cleft lip repairs, non-head injuries such as fractures, drainage of subungual or perichondrial haematomata).
- relatives: Any familly members of included patient, aged of 2 or more. Exept persons with profound intellectual disability

SUMMARY:
The main objective of the study is to define, for Autism Spectrum Disorder, the extent of genetic variation in synaptic pathways that may be targeted for therapeutic development. For this purpose the investigators will take advantage of large, well-characterized cohorts of patients with Autism Spectrum Disorder for genetic screenings. Targeted sequencing of selected synaptic genes, previously associated with Autism Spectrum Disorder, will be carried out in these cohorts with deep coverage of coding regions and a strong focus on previously untested regulatory regions. Genomic data from Copy Number Variant, whole genome sequencing and exome sequencing, available for some of these patients, will be integrated in the overall analysis. The investigators will strongly emphasize the establishment of comprehensive genotype/phenotype correlations and set up an induced Pluripotent Stem Cells collection from selected patients with synaptic mutations for functional and expression analysis.

DETAILED DESCRIPTION:
Specific aims are:

Aim 1: To identify genetic variants in selected synaptic genes, by targeted sequencing with deep coverage of coding regions and a strong focus on previously untested regulatory regions in Autism Spectrum Disorder

Aim 2: To define the range of clinical phenotypes caused by mutations in synaptic genes by establishing detailed genotype/phenotype correlations and analyzing segregation in families with multiple individuals affected by Autism Spectrum Disorder, Autism Spectrum Disorder traits or other neuropsychiatric disorders

Aim 3: To generate a repository of induced Pluripotent Stem Cells from Autism Spectrum Disorder subjects with synaptic mutations for translational studies, including expression and functional assays.

Aim 4: To identify the neuronal phenotypes caused by deleterious synaptic mutations for further translational studies

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis for Autism Spectrum Disorders or Autism using the Autism Diagnostic Interview-Revised (ADI-R) criteria for autism and Autism Diagnostic Observation Schedule (ADOS-G) criteria

Exclusion Criteria:

* Patients with profound intellectual disability or with a known medical cause of autism, such as neurocutaneous syndromes, Fragile X, metabolic disorders, extreme prematurity, congenital rubella and other prenatal or postnatal neurological infections or gross dysmorphology, will be excluded

Ages: 18 Months to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For all patients included in the study, .
Sampling Method: Non-Probability Sample
Enrollment: 1616 (Actual)
Dates: Start 2009-02-04 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of synaptic gene deleterious mutations in patients with Autism Spectrum Disorder | up to 12 months after completion of the inclusion and molecular explorations

SECONDARY OUTCOMES:
Prevalence of the deleterious mutations in the major biological pathways in Autism Spectrum Disorders: | up to 12 months after completion of the inclusion and molecular explorations)
  The deleterious mutations that the investigators will identify in genes related to Autism Spectrum Disorders will help to have a comprehensive framework of biological pathways involved in Autism Spectrum Disorder

CONTACTS AND LOCATIONS:
Overall Officials: Marion Leboyer, M.D, Ph.D, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (5):
- France (5):
  - Centre de Ressources Autisme Aquitaine, CHU de Bordeaux, Bordeaux
  - CADIPA Centree hospitalier de Saint Egreve, Grenoble
  - Cic Henri Mondor, Paris
  - Albert Chenevier Hospital, Créteil, Île-de-France Region
  - Robert Debré Hospital, Paris, Île-de-France Region

REFERENCES:
- [Background] Delorme R, Ey E, Toro R, Leboyer M, Gillberg C, Bourgeron T. Progress toward treatments for synaptic defects in autism. Nat Med. 2013 Jun;19(6):685-94. doi: 10.1038/nm.3193. Epub 2013 Jun 6. PMID 23744158
- [Derived] Amestoy A, Guillaud E, Bucchioni G, Zalla T, Umbricht D, Chatham C, Murtagh L, Houenou J, Delorme R, Moal ML, Leboyer M, Bouvard M, Cazalets JR. Visual attention and inhibitory control in children, teenagers and adults with autism without intellectual disability: results of oculomotor tasks from a 2-year longitudinal follow-up study (InFoR). Mol Autism. 2021 Nov 13;12(1):71. doi: 10.1186/s13229-021-00474-2. PMID 34774105
- [Derived] Latimier A, Kovarski K, Peyre H, Fernandez LG, Gras D, Leboyer M, Zalla T. Trustworthiness and Dominance Personality Traits' Judgments in Adults with Autism Spectrum Disorder. J Autism Dev Disord. 2019 Nov;49(11):4535-4546. doi: 10.1007/s10803-019-04163-1. PMID 31418129
- [Derived] Grea H, Scheid I, Gaman A, Rogemond V, Gillet S, Honnorat J, Bolognani F, Czech C, Bouquet C, Toledano E, Bouvard M, Delorme R, Groc L, Leboyer M. Clinical and autoimmune features of a patient with autism spectrum disorder seropositive for anti-NMDA-receptor autoantibody. Dialogues Clin Neurosci. 2017 Mar;19(1):65-70. doi: 10.31887/DCNS.2017.19.1/mleboyer. PMID 28566948
- See also: website of the sponsor — http://www.inserm.fr
- See also: Site de transparence — https://www.fondation-fondamental.org/faire-avancer-la-recherche/les-projets-de-fondamental/projet-genes-et-autisme